CLINICAL TRIAL: NCT01124136
Title: Evaluation of the Effect of Neurostimulation in Patients With Symptomatic Heart Failure
Brief Title: Neurostimulation of Spinal Nerves That Affect the Heart
Acronym: Neurostim
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jerry Estep, MD (Other)
Collaborators: The Methodist Hospital Research Institute (Other)
Responsible Party: Sponsor-Investigator, Jerry Estep, MD, Sponsor-Investigator/Principal Investigator, The Methodist Hospital Research Institute
Organization: The Methodist Hospital Research Institute (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00002132; 0708-0211 (Other: HMRI IRB)
Record Dates: First submitted 2010-05-10; First posted 2010-05-14 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Chronic Heart Failure
Keywords: Chronic Heart Failure; Neurostimulation
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Heart failure treatment standard of care (SOC) consists of medication management to support heart and manage symptoms. In this study, patients will receive the neurostimulator + SOC or SOC only.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Neurostimulation + Medication management (Experimental): Investigational nerve stimulator device implanted to heart plus standard medication therapy.
  Interventions: Device: Neurostimulation + Medication Management (Standard of Care); Drug: Standard of Care (Control)
- Standard of Care (Control) (Other): Standard of Care treatment is medication management only. Heart failure medications control symptoms and comorbidities, i.e. blood thinners, lipid lowering, and diuretics, and manage heart function, i.e. heart rhythm, rate, and pumping strength.
  Interventions: Drug: Standard of Care (Control)

INTERVENTIONS:
Device: Neurostimulation + Medication Management (Standard of Care) — In addition to medication management, adding investigational implanted neurostimulator to heart
  Other Names: Neurostimulator and medication management
  Arms: Neurostimulation + Medication management
Drug: Standard of Care (Control) — Standard of Care Therapy consists of medication management only to support heart for rhythm, anticoagulation, and rate, and comorbid symptoms, i.e. diuretics, lipid lowering.
  Other Names: Standard Care, Medical Management only

SUMMARY:
The purpose of this study is to study the use of neurostimulation in chronic advanced refractory heart failure.

The study is determine if it is safe to use neurostimulation in patients with chronic advanced refractory heart failure and to also determine initial observations with regards to its potential effect on heart function and quality of life. The investigators hypothesis is that this study will show both safe and positive effect of neurostimulation on heart failure patients.

DETAILED DESCRIPTION:
Protocol Summary

Title EVALUATION OF THE SAFETY OF NEUROSTIMULATION IN PATIENTS WITH SYMPTOMATIC HEART FAILURE FEASIBILTIY STUDY

Description A feasibility trial of the use of neurostimulation in chronic advanced refractory heart failure.

Objective To determine the safety of neurostimulation in patients with chronic advanced refractory heart failure and to generate initial observations with regards to its potential effect on ventricular function and quality of life.

Design The trial will be a randomized double blind crossover feasibility trial with 2 week and 1,2,3,4,5,6,7 month clinical follow-up.

After device implantation, patients enrolled in the trial will have been randomly assigned to have device programmed to deliver impulses, active, or to have the device programmed not to deliver impulses, inactive, for 3 months.

After the 3 month initial phase, the devices will be inactivated and a 4 week washout period will convene.

At the end of washout period, patients that were inactive during initial phase will crossover to active and similarly patients that were active during initial phase will crossover to inactive.

Patient Population Patients with non-ischemic or ischemic cardiomyopathy with a length of illness of at least 6 months who have met the inclusion and exclusion criteria.

Enrollment Enrollment of a total of 10 intent-to-treat patients Investigational Sites Up to 2 investigational sites in the US Data Collection Data collection will be obtained in three categories: markers of cardiovascular safety, markers of device-device interactions and markers of efficacy.

ELIGIBILITY:
Inclusion

1. Male or female ≥18 years;
2. Chronic heart failure NYHA class III-IV of ischemic and non-ischemic etiology;
3. Screening Left ventricular Ejection Fraction (LVEF) ≤ 30% measured at baseline by echocardiography;
4. Screening 6 minute walk test score of less than 450 meters measured at baseline;
5. Hospitalization for heart failure or outpatient IV administration of inotropic agents, human B-natriuretic peptide or IV diuretics within the past 12 months (stable for at least 2 weeks);
6. On standard optimal medical therapy for CHF before medical therapy.*
7. No changes in active cardiac medications during the 1 week prior to treatment;
8. Written informed consent.

   * Patients with current or prior symptoms of heart failure and reduced LVEF should be on stable optimally uptitrated medical therapy recommended according to current guidelines (Circulation. 2005; 112 (12): e154) as standard of care for heart failure therapy in the United States. This minimally includes an ACE-inhibitor (ACE-I) at stable doses for 1 month prior to enrollment, if tolerated, and a beta blocker (carvedilol, metoprolol succinate, or bisoprolol) for 3 months prior to enrollment, if tolerated, with a stable up-titrated dose for 1 month prior to enrollment. This also includes an Angiotensin II Receptor Blocker (ARB) at stable doses for 1 month prior to enrollment, if tolerated, when ACE-I is not tolerated. Stable is defined as no more than a 100% increase or a 50% decrease in dose. If the patient is intolerant to ACE-I, ARB, or beta blockers, documented evidence must be available. In those intolerant to both ACE-I and ARB, combination therapy with hydralazine and oral nitrate should be considered. Therapeutic equivalence for ACE-I substitutions is allowed within the enrollment stability timelines. Aldosterone inhibitor therapy should be added when NYHA Class III or IV symptoms occur on standard therapy. If aldosterone inhibitor therapy is administered in Class II patients, it must be initiated and optimized prior to enrollment. Eplerenone requires dosage stability for 1 month prior to enrollment. Diuretics may be used as necessary to keep the patient euvolemic.

Exclusion

1. Inability to comply with the conditions of the protocol;
2. Inability to perform cardiopulmonary exercise test due to mechanical physical limitations
3. Presence of a transplanted tissue or organ or LVAD (or the expectation of the same within the next 12 months);
4. Planned AICD or CRT within the next 12 months unless AICD is prescribed for primary prevention
5. Pacemaker dependent patients.
6. Acute MI, CABG, PTCA, within the past 3 months
7. Chronic refractory angina or peripheral vascular pain;
8. Valvular heart disease requiring repair or replacement;
9. Need for chronic intermittent inotropic therapy;
10. Malignancy: evidence of disease within the previous 5 years;
11. Known HIV infection or immunodeficiency state;
12. Chronic active viral infection (such as hepatitis B or C);
13. Severe systemic infection: defined as patients undergoing treatment with antibiotics;
14. Active myocarditis or early postpartum cardiomyopathy (within the first 6-months of delivery);
15. Systemic corticosteroids, cytostatics and immunosuppressive drug therapy (cyclophosphamide, methotrexate, cyclosporine, azathioprine, etc.), DNA depleting or cytotoxic drugs taken within 4 weeks prior to study treatment;
16. Patient is pregnant, of childbearing potential and not using adequate contraceptive methods, or nursing.;
17. Patient scheduled for hospice care;
18. Any other medical, social or geographical factor, which would make it unlikely that the patient will comply with study procedures (eg. Alcohol abuse, lack of permanent residence, severe depression, disorientation, distant location and a history of non-compliance).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-05; Primary Completion 2018-10 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Markers of cardiovascular safety | 2 years
  Markers of cardiovascular safety will include specific clinical events that define worsening of heart failure including hospitalization for worsening heart failure, symptomatic brady-arrhythmia or tachy-arrhythmia necessitating cardioversion or death.
Markers of device-device interaction | 2 years
  Markers of device-device interaction will include failure to properly provide pacing or adequate defibrillation or inappropriate shocks. Also, failure to initiate neurostimluation as programmed by the protocol
Markers of efficacy | Average: till the end of the study
  Markers of efficacy will include change in left ventricular ejection fraction as determined by echocardiography, change in maximal oxygen consumption as measured by cardio-pulmonary exercise testing, and change in quality of life as measured by the MLHFQ. Other exploratory markers include measurements in diastolic function by echocardiography, changes in neurohormonal and inflammatory markers, specifically BNP, plasma cytokines(TNF alpha and IL 6), complement, and C-reactive protein.

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Estep, MD, Principal Investigator — Methodist Hospital DeBakey Heart & Vascular Center
Locations (1):
- Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
to be determined